CLINICAL TRIAL: NCT01546415
Title: A Single Arm, Multicenter, Open Label Study of Desferasirox in Chinese Patients With Iron Overload and Aplastic Anemia
Brief Title: Safety and Efficacy of Desferasirox in Chinese Patients With Iron Overload and Aplastic Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ACN01
Record Dates: First submitted 2011-11-10; First posted 2012-03-07 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Iron Overload
Keywords: Phase 4; Desferasirox; Iron Overload; Aplastic Anemia
MeSH Terms: conditions — Iron Overload; Anemia, Aplastic

ARMS (1):
- Desferasirox (Experimental)
  Interventions: Drug: Desferasirox

INTERVENTIONS:
Drug: Desferasirox — Initial Dose: 20 mg/kg/d. Dose modification according to protocol.

SUMMARY:
The study is designed to collect safety and efficacy of Desferasirox in Chinese patients with Iron Overload and Aplastic Anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with transfusion-related IOL as shown by a SF level of ≥ 1000 ng/mL at start of study
* History of transfusion >20 international units or 100 mL/kg of red blood cells
* Underlying transfusion-dependent illness:

  * AA: Clinically diagnosed AA with bone marrow confirmation of the diagnosis
* Age ≥ 18 years, male or female
* Written informed consent obtained from patient prior to any screening procedures.

Exclusion Criteria:

* Patients with serum creatinine > ULN or with significant proteinuria as indicated by a urinary protein/creatinine ratio (UPCR) ≥ 1.0 mg/mg in a non-first void urine sample at baseline. If serum creatinine is found to be > ULN or UPCR is found to be ≥ 1 mg/mg the test can be repeated after 1 month.
* Creatinine Clearance <40 ml/min
* Patients with other than AA transfusion-dependent underlying illnesses
* Patients with a previous history of clinically relevant ocular and/or auditory toxicity related to iron chelation
* Any other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug. The investigator should be guided by evidence of any of the following:
* history of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding
* history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
* history of pancreatic injury or pancreatitis; indications of impaired pancreatic function/injury as indicated by abnormal lipase or amylase
* history or presence of impaired renal function as indicated by creatinine or blood urea nitrogen (BUN) values equal or above ULN
* history of urinary obstruction or difficulty in voiding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in serum ferritin from baseline to 52 weeks with desferasirox treatment in Chinese patients with AA presenting with transfusional hemosiderosis and pre-existing serum ferritin levels of ≥ 1000 ng/mL. | Every 4 Weeks for 52 weeks of treatment
  Difference in serum ferritin from baseline vs. 52 weeks of treatment.

SECONDARY OUTCOMES:
Correlation between serum ferritin (SF) and transferrin saturation (TFS) | Every 4 Weeks for 52 weeks of treatment
  Study will compare SF with TFS level to find degree of relationship measured by correlation.
Number of dispensed, used, partially used or unused packages of study medication to assess drug usage compliance | Every 4 Weeks for 52 weeks of treatment
Correlation between dose adjustment (increase or decrease) regimens and transfusional burden | Every 3 months for 52 Weeks of treatment
  Evaluation of the relationship between dose adjustment regimens (as dictated by both efficacy and safety parameters) and transfusional burden will be undertaken.
Number of patients with adverse events, serious adverse events and death | Every 4 weeks for 52 Weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- China (7):
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chengdu
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin

REFERENCES:
- [Derived] Shi J, Chang H, Zhang L, Shao Y, Nie N, Zhang J, Huang J, Zhang L, Tang X, Quan R, Zheng C, Xiao H, Hu D, Hu L, Liu F, Zhou Y, Zheng Y, Zhang F. [Efficacy and safety of deferasirox in aplastic anemia patients with iron overload: a single arm, multi-center,prospective study in China]. Zhonghua Xue Ye Xue Za Zhi. 2016 Jan;37(1):1-6. doi: 10.3760/cma.j.issn.0253-2727.2016.01.001. Chinese. PMID 26876245